CLINICAL TRIAL: NCT02156115
Title: Characterization of the Pathogenesis of Primary and Secondary Lymphatic Disorders
Status: Terminated | Type: Observational
Why Stopped: Study closed before total enrollment met.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 140127; 14-H-0127
Record Dates: First submitted 2014-06-04; First posted 2014-06-05 (Estimated); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Lymphangiomatosis; Lymphedema; Lymphangiectasia; Pulmonary Lymphangiectasia
Keywords: Lymphangiomatosis; Lymphangiogenesis; Smooth Muscle Cell; Vascular Anomalies; Natural History
MeSH Terms: conditions — Lymphedema; Lymphangiectasis; Vascular Malformations

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy volunteers: healthy volunteers
- lymphatic patients: lymphatic patients
- relatives: relatives

SUMMARY:
Background:

- Lymphatics are a type of vessel, similar to arteries and veins. Lymphatic disorders happen when these vessels don t work properly. Researchers want to look for a relationship between lymphatic disorders and variations of certain genes found in the lung, blood, and other places in the body.

Objective:

- To learn more about lymphatic disorders and evaluate how genetic factors affect lymphatic disorders.

Eligibility:

* People ages 2 90 who have a lymphatic disorder or relatives of people with lymphatic disorders.
* Healthy volunteers 18 and older.

Design:

* Participants may have 1 2 visits a year, or more as needed. The study is expected to last 5 years. Visits may last 1 5 days. Participants may have lab tests, medical history, and physical exam at each visit.
* Participants may have blood testing that includes genetics tests, and urine tests. They may have nose and throat cultures, saliva collection, and cheek swabs to collect samples.
* Participants may have a skin biopsy and have blood taken from an artery.
* Participants may have breathing tests and be studied while exercising.
* Participants may have an electrocardiogram. Electrodes will be placed on their chest, tracing heart rhythms. They may also have chest X-rays.
* Participants may have a bronchoscopy. A thin, flexible instrument will be passed through the nose or mouth, into the lung. A tissue sample will be taken.
* Participants who have lymphatic disease or have a relative with it may also have:
* CT scans. They will lie on a table and hold their breath while their chest is scanned.
* MRI. They will lie flat on a table that slides in and out of a scanner.
* ultrasound. A probe is rolled around outside the abdomen.
* removal of fluid around the lungs, chest, and abdomen.

DETAILED DESCRIPTION:
Disorders of lymphatic function are associated with multiple presentations, the most common of which is lymphedema, a chronic swelling of the extremities, due to impaired lymphatic drainage. It can cause disability and a predisposition to infection and chronic ulceration. Other lymphatic disorders present with visceral manifestations such as regional or systemic lymphangiomatosis, pulmonary and intestinal lymphangiectasia, protein-losing enteropathy, chylous ascites, and chylothorax. Abnormalities of smooth muscle cell proliferation are associated with lymphangiomatosis. Proliferation of a neoplastic cell, the LAM cell, which exhibits a smooth muscle cell phenotype, is associated with lymphangioleiomyomatosis. Currently, treatment for many of these disorders is symptomatic and the prognosis is variable.

The molecular mechanisms of lymphatic vasculogenesis are incompletely understood, but critical genes have been described, and mutations in these genes may lead to developmental abnormalities. There may be a genetic predisposition to lymphatic disorders, with a role for modifier genes in disease progression. The purpose of this study is to (a) define the natural history of lymphatic diseases, (b) characterize the clinical phenotypes, and (c) elucidate their pathogenesis at the physiological, cellular and molecular levels. This protocol is part of a Trans-Institute basic, translational and clinical initiative in lymphatic disorders and will include participation of principal investigators across the NIH, as well as extramural investigators.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Patients 2 years of age or older with clinical or histological evidence for a lymphatic abnormality; patients will in the vast majority of cases be referred with the diagnosis of a lymphatic disorder.
  2. Patients 2 years of age or older with findings on physical examination consistent with the diagnosis of a lymphatic abnormality.
  3. Relatives of patients with lymphatic disorders, 2 years of age or older.
  4. Healthy research volunteers 18 years of age or older as control subjects.

EXCLUSION CRITERIA:

1. Patients who are less than 2 years of age. Research volunteers less than 18 years of age. Age greater than 90 years old.
2. Advanced stage of any systemic illness.
3. An exclusion criterion for participating in the x-ray portion of the study is pregnancy.
4. Exclusion criteria for participating in the bronchoscopy portion of the study are: (1) presence of any contraindication for fiberoptic bronchoscopy, with lavage and/or bronchial brushing; (2) advanced stage of a pulmonary or a systemic illness such that the risk is judged to be significant even in the absence of a specific contraindication to the procedure; (3) allergy to topical anesthetic (e. g., lidocaine); (4) current or recent respiratory infection (within the last 4 weeks); (5) pregnancy or lactation; (6) age less than 18 or greater than 65.
5. Exclusion criteria for participating in the endoscopy portion of the study are: (1) Any medical, psychiatric, or social conditions which, in the opinion of the investigators, would make participation in this protocol not in the best interest of the patient; (2) have a history of surgical removal of a portion or all of the colon if it is believed to increase risk; (3) are pregnant; (4) have had radiation to the abdomen or pelvis; (5) have poor heart or lung function that would make sedation too risky; (6) have allergy or other contraindications to midazolam or fentanyl; (7) are unable to tolerate preparation for the procedure; (8) are unable to give consent; (9) have had abdominal surgery within eight weeks; (10) are taking anticoagulant therapy that cannot be interrupted; (11) have had diverticulitis or an abdominal abscess within eight weeks.

Ages: 2 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include any individual 2 years of age or older with definite or probable diagnosis of a lymphatic disorder and age, race and sex matched healthy volunteers as a control group for patients 18 years of age and above. Relatives of individuals with lymphatic disorders are also eligible for participation.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
(a) define the natural history of lymphatic diseases, (b) characterize the clinical phenotypes, and (c) elucidate their pathogenesis at the physiological, cellular and molecular levels. | ongoing
  To define the clinical phenotype of the lymphatic disorder.To define the molecular basis of the lymphatic disorders.This knowledge will help in improving our understanding of lymphatic proliferation in normal conditions as well as in disease.

SECONDARY OUTCOMES:
To assess the contribution of proteins and other genes to the clinical phenotype. | Undefined

CONTACTS AND LOCATIONS:
Overall Officials: Joel Moss, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2014-H-0127.html